CLINICAL TRIAL: NCT02598895
Title: Docetaxel and Carboplatin for Patients With Metastatic, Castration Resistant Prostate Cancer and Inactivated Genes in BRCA 1/2 Pathway
Brief Title: Docetaxel and Carboplatin in Treating Patients With Metastatic, Castration Resistant Prostate Cancer Containing Inactivated Genes in the BRCA 1/2 Pathway
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Cheng, Associate Professor, University of Washington, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9381; NCI-2015-01694 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9381 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); P50CA097186 (NIH); RG1715099 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-10-13; First posted 2015-11-06 (Estimated); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; PSA Progression; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (docetaxel, carboplatin) (Experimental): Patients receive docetaxel IV over 30-60 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies docetaxel and carboplatin in treating patients with castration resistant prostate cancer that has spread from the primary site (place where it started) to other places in the body (metastatic) and contains inactivated genes in the BRCA 1/2 pathway. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive docetaxel intravenously (IV) over 30-60 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 10 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information
* Histologically or cytologically confirmed carcinoma of the prostate (excluding neuroendocrine differentiation or squamous cell histology)
* Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy; patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy
* Castration resistant prostate cancer as defined by rising PSA when serum testosterone < 50 ng/ml (note: current testosterone results are not required if the potential subject has not missed any GnRH analogue/antagonist doses since their last result was received) AND one of the following:

  * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
  * Evaluable disease progression by modified RECIST (Response Evaluation Criteria in Solid Tumors)
  * Progression of metastatic bone disease on bone scan with > 2 new lesions
* Prior therapy with abiraterone, enzalutamide and/or docetaxel; there is no limit to the number of prior treatment regimens
* Presence of metastatic disease on scans
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy >= 12 weeks
* No prior malignancy is allowed except:

  * Adequately treated basal cell or squamous cell skin cancer or
  * In situ carcinoma of any site or
  * Other adequately treated malignancy for which the patient has been disease-free for at least one year (any prior chemotherapy is allowed)
* Absolute neutrophil count >= 1.5 x 10^9 cells/L
* Hemoglobin (Hgb) >= 9.0 g/dL
* Platelets >= 100,000 x 10^9/L
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN)
* Total bilirubin levels =< 1.5 x ULN
* Patients must have clear and documented evidence of biallelic inactivation BRCA1, BRCA2 or ATM by sequencing, for example University of Washington (UW)-Oncoplex, SU2C, or Foundation One testing and/or patients with clearly deleterious mutations of other genes involved in homologous DNA repair (e.g., partner and localizer of BRCA2 [PALB2], BRCA1-interacting protein 1 [BRIP1], etc.) by sequencing via UW-Oncoplex, SU2C, or Foundation One testing may be included at the investigator's discretion

Exclusion Criteria:

* Currently receiving active therapy for other neoplastic disorders
* Histologic evidence of neuroendocrine or small cell carcinoma of the prostate
* Known parenchymal brain metastasis
* Active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease or cardiac ejection fraction measurement of < 35 % at baseline, if done
* Treatment with an investigational therapeutic within 30 days of cycle 1
* Patients with dementia/psychiatric illness/social situations limiting compliance with study requirements or understanding and/or giving of informed consent are not eligible
* Any medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained are not eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather H. Cheng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Docetaxel, Carboplatin)
Started | 14
PSA50 | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Docetaxel, Carboplatin)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] — Age in years at enrollment
  years | 64 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With PSA Decline by 50% From Baseline
Description: Proportion of patients with PSA decline by 50% from baseline according to Prostate Cancer Working Group 2 (PCWG2) criteria
Time Frame: Until disease progression or unacceptable toxicity, assessed up to 35 days after the last dose of study medication
Population: Patients treated with docetaxel and carboplatin.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Docetaxel, Carboplatin)
Number analyzed (Participants) | 14
Participants
  achieved PSA50 | 9
  did not achieve PSA50 | 5
Statistical Analysis 1: Comparison: Treatment (Docetaxel, Carboplatin); The primary efficacy endpoint was percent patients achieving PSA decline of 50% or more from baseline (PSA50), assessed in the time prior to disease progression, unacceptable toxicity or 1 year after the last study medication. The historical comparison was PSA50 of 26%. The target response rate was 60%. The study followed an optimal two-stage Simon design (Simon, 1989) where the null hypothesis that the true PSA response rate PSA50 was 0.26 was tested against a one-sided alternative; Test type: Other; See above

ADVERSE EVENTS:
Time Frame: Adverse events data were collected up to 2.5 years after the last dose of study treatment for each participant.
Description: The investigator was responsible for ensuring that all non-serious grade 3 and above non-serious adverse events (as defined in Section 6.7.1 and as further specified below) observed by the investigator or reported by subjects were collected and recorded in the CRF. Source documents may have included the subjects' medical records, patient diaries or study-specific worksheets. Recording for all events were done in a concise manner using standard, acceptable medical terms.
Arm/Group | Treatment (Docetaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 10/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Docetaxel, Carboplatin) (N=14)
Platelet Count Decreased (Blood and lymphatic system disorders) | 4 (9) — Platelet Count Decreased
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1 (1) — Neutropenia
Anemia (Blood and lymphatic system disorders) | 2 (2) — Anemia
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT02598895/Prot_SAP_000.pdf